CLINICAL TRIAL: NCT03613103
Title: Airway Injuries After Intubation Using Videolaryngoscopy Highly Curved Blades Versus Direct Laryngoscopy for Adult Patients Requiring Tracheal Intubation: a Randomized Controlled Trial
Brief Title: Airway Injuries After Intubation Using Videolaryngoscopy Versus Direct Laryngoscopy for Adult Patients Requiring Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: IPS Universitaria-Universidad de Antioquia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Airway - 001
Record Dates: First submitted 2018-07-03; First posted 2018-08-02 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Airway Trauma; Airway Complication of Anesthesia
Keywords: video laryngoscopy; airway; injury; direct laryngoscopy; intubation; endotracheal
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A single-center randomized study is performed including non-cardiac surgical patients without predictable risk of difficult mask ventilation or of difficult tracheal intubation. For direct laryngoscopy group, we use a Macintosh blade and for videolaryngoscopy group we use videolaryngoscopy highly curved blade. Induction of anesthesia is performed using myorelaxation with rocuronium. We record each five minute the vital signs in the anesthesia record. The primary outcome is observed injuries in the mucosa of the airway: Erythema, edema, ecchymosis, laceration, excoriation and / or hematoma. Injuries to dental pieces: Partial and / or total loss of tooth integrity, loosening of dental piece, damage to dental and / or aesthetic prosthetic material. Laryngeal lesions: Edema, laceration, excoriation, erythema, ecchymosis and / or bleeding pharyngeal laryngeal mucosa, arytenoid luxation. Post-intubation symptoms: Sore throat, dysphonia and / or aphonia.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned at the time of anesthetic induction in the surgery room. The allocation to the direct laryngoscopy group and the video laryngoscopy will be 1: 1 randomly using permuted blocks, generated by a computer operated by an external assistant to the investigation. The size of the blocks will be between 4, 6, and 8.
  A person external to the research group will be responsible for concealment of allocation through opaque and sealed envelopes, listed sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct laryngoscopy (Active Comparator): Intubation with direct laryngoscopy (Conventional Intubation)
  Interventions: Device: Direct laryngoscopy
- Videolaryngoscopy (Experimental): Intubation with videolaryngoscopy (Assisted video intubation)
  Interventions: Device: Video laryngoscopy

INTERVENTIONS:
Device: Video laryngoscopy — Intubation with videolaryngoscopy with highly curved blade
  Arms: Videolaryngoscopy
Device: Direct laryngoscopy — Intubation with direct laryngoscopy with macintosh blade
  Arms: Direct laryngoscopy

SUMMARY:
Abstract Background Successful tracheal intubation during general anesthesia requires a direct laryngoscope to retract the tongue and soft tissues of the mouth to achieve a line of sight for the larynx. Generally, Macintosh blade laryngoscopy is used to achieve the tracheal intubation. However, difficulties with the tracheal intubation arise the need to use alternative laryngoscopes that use digital or fiberoptic technology, to improve the larynx visibility. Among these devices, highly curved blade videolaryngoscope uses a curved blade to retract the soft tissues of floor of the mouth and transmits a video image to a screen, achieving better larynx visibility. Also, the decrease of the force in the soft tissues with videolaryngoscope could reduce airway injures.

Objectives Our primary objective is to assess whether use of videolaryngoscopy using highly curved blades for tracheal intubation in adults requiring general anesthesia reduces risk of airways injuries compared with Macintosh direct laryngoscopy. Our secondary aim is to assess postoperative satisfaction of the patients, successful intubation at the first attempt, successful global intubation, degree of larynx visibility according to classification Cormack - Lehane and time taken to perform intubation in videolaryngoscopy vs direct laryngoscopy. Finally, we assess the risk of presenting serious adverse event with the use of videolaryngoscopy compared with Macintosh laryngoscopy in hypoxemia, bradycardia and heart arrest.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Scheduled for a procedure or surgery that requires general anesthesia that requires orotracheal intubation.
* Scheduled for non-cardiac surgery.
* Elective surgery.

Exclusion Criteria:

* Women in pregnancy.
* Patient refuses to participate in the study before surgery.
* Patients with predictors of anticipated difficult airway.
* Head and neck surgery.
* Go to Intensive Care Unit with endotracheal intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an airway injury | 24 hours
  Airway injury will be a composite outcome as follow: Injury in the oral cavity or injury in the laryngopharynx.
  These injuries will be evaluated using a digital camera of the oral cavity (fiber optical camera) in the immediate POP.
  A patient will be considered positive for the outcome If he/she has at least one of the following findings: Erythema, edema, ecchymosis, laceration, excoriation and / or hematoma in labial, jugal, gingival, lingual mucosa, hard and soft palate; Dental pieces injury: partial and / or total loss of the integrity of the dental piece; Larynx lesions: Edema, laceration, excoriation, erythema, ecchymosis and / or bleeding of pharyngeal laryngeal mucosa.

SECONDARY OUTCOMES:
Successful intubation at the first attempt | Immediate postoperative
  Number of patients with successful intubation at the first attempt.
Global of Successful Intubation | Immediate postoperative
  Number of patients with successful intubation regardless of the attempts to achieve it.
Cormack-lehane visualization | Immediate postoperative
  Degree of Cormack-lehane visualization in each patient. The degree of Cormack-Lehane visualization will be measured from I to IV in relation to the visible portion of the glottis; Grade I with total visualization and Grade IV without visualization of glottis.
Time to achieve orotracheal intubation | Immediate postoperative
  Time measured in seconds to achieve orotracheal intubation in each patient. The time interval is determined from the beginning of laryngoscopy by the anesthesiologist until the verification of tracheal intubation by capnography.
Post-anesthetic satisfaction | Immediate postoperative
  Post-anesthetic satisfaction in each patient. The Quality of Recovery scale 40 will be used to determine the degree of patient satisfaction, according to the overall and subglobal score, defined by five dimensions: patient support, comfort, emotional, physical independence and pain (includes anatomical airway site).
Hypoxemia during induction and intubation | Immediate postoperative
  Number of patients with hypoxemia during induction and intubation. Hypoxaemia is defined as an oxygen saturation measured with pulse oximetry less than 92%.
Bradycardia during induction and intubation | Immediate postoperative
  Number of patients with bradycardia during induction and intubation. Bradycardia is defined as a decrease in heart rate of less than 40 beats / minute.
Cardiac Arrest | Immediate postoperative
  Number of patients presenting cardiac arrest. Cardiac arrest is defined as the presence of any malignant rhythm: Ventricular tachycardia, ventricular fibrillation, asystole or pulseless electrical activity plus loss of carotid pulse for more than 10 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonathan Benumof CAH. Benumof and Hagberg's Airway Management - Jonathan Benumof, Carin A. Hagberg [Internet]. Third Edit. Carin A. Hagberg (The University of Texas MS at H, editor. Elsevier. Philadelphia, PA 19103-2899: Elsevier Inc; 2013. 1142 p. Available from: www.elsevier.com/permissions.
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Scott J, Baker PA. How did the Macintosh laryngoscope become so popular? Paediatr Anaesth. 2009 Jul;19 Suppl 1:24-9. doi: 10.1111/j.1460-9592.2009.03026.x. PMID 19572841
- [Background] Abeyewardene L, Ganta R, Henthorn R. Direct laryngoscopy with the aid of a fiberoptic bronchoscope for tracheal intubation. Anesth Analg. 1996 Sep;83(3):665. doi: 10.1097/00000539-199609000-00066. No abstract available. PMID 8780318
- [Background] Parasa M, Yallapragada SV, Vemuri NN, Shaik MS. Comparison of GlideScope video laryngoscope with Macintosh laryngoscope in adult patients undergoing elective surgical procedures. Anesth Essays Res. 2016 May-Aug;10(2):245-9. doi: 10.4103/0259-1162.167840. PMID 27212755
- [Background] De Jong A, Molinari N, Conseil M, Coisel Y, Pouzeratte Y, Belafia F, Jung B, Chanques G, Jaber S. Video laryngoscopy versus direct laryngoscopy for orotracheal intubation in the intensive care unit: a systematic review and meta-analysis. Intensive Care Med. 2014 May;40(5):629-39. doi: 10.1007/s00134-014-3236-5. Epub 2014 Feb 21. PMID 24556912
- [Background] Kaplan MB, Ward DS, Berci G. A new video laryngoscope-an aid to intubation and teaching. J Clin Anesth. 2002 Dec;14(8):620-6. doi: 10.1016/s0952-8180(02)00457-9. PMID 12565125
- [Background] Jarvis JL, McClure SF, Johns D. EMS Intubation Improves with King Vision Video Laryngoscopy. Prehosp Emerg Care. 2015;19(4):482-9. doi: 10.3109/10903127.2015.1005259. Epub 2015 Apr 24. PMID 25909850
- [Background] Lu Y, Jiang H, Zhu YS. Airtraq laryngoscope versus conventional Macintosh laryngoscope: a systematic review and meta-analysis. Anaesthesia. 2011 Dec;66(12):1160-7. doi: 10.1111/j.1365-2044.2011.06871.x. Epub 2011 Aug 25. PMID 21883130
- [Background] Turkstra TP, Pelz DM, Jones PM. Cervical spine motion: a fluoroscopic comparison of the AirTraq Laryngoscope versus the Macintosh laryngoscope. Anesthesiology. 2009 Jul;111(1):97-101. doi: 10.1097/ALN.0b013e3181a8649f. PMID 19512871
- [Background] Kill C, Risse J, Wallot P, Seidl P, Steinfeldt T, Wulf H. Videolaryngoscopy with glidescope reduces cervical spine movement in patients with unsecured cervical spine. J Emerg Med. 2013 Apr;44(4):750-6. doi: 10.1016/j.jemermed.2012.07.080. Epub 2013 Jan 22. PMID 23351572
- [Background] Kramer A, Muller D, Pfortner R, Mohr C, Groeben H. Fibreoptic vs videolaryngoscopic (C-MAC((R)) D-BLADE) nasal awake intubation under local anaesthesia. Anaesthesia. 2015 Apr;70(4):400-6. doi: 10.1111/anae.13016. PMID 25764403
- [Background] Hunter I, Ramanathan V, Balasubramanian P, Evans DA, Hardman JG, McCahon RA. Retention of laryngoscopy skills in medical students: a randomised, cross-over study of the Macintosh, A.P. Advance() , C-MAC((R)) and Airtraq((R)) laryngoscopes. Anaesthesia. 2016 Oct;71(10):1191-7. doi: 10.1111/anae.13589. Epub 2016 Aug 17. PMID 27530359
- [Background] Graham B. Defining and Measuring Patient Satisfaction. J Hand Surg Am. 2016 Sep;41(9):929-31. doi: 10.1016/j.jhsa.2016.07.109. PMID 27570227
- [Background] Castellanos-Olivares DA, Evangelina-Cervantes DH, Vásquez-Márquez DPI. Satisfacción anestésica como indicador de calidad de la atención médica en el paciente geriátrico. Rev Mex Anestesiol [Internet]. 2013;36(1):250-5. Available from: /www.medigraphic.com/pdfs/rma/cma-2013/cmas131be.pdf
- [Background] Barnett SF, Alagar RK, Grocott MP, Giannaris S, Dick JR, Moonesinghe SR. Patient-satisfaction measures in anesthesia: qualitative systematic review. Anesthesiology. 2013 Aug;119(2):452-78. doi: 10.1097/ALN.0b013e3182976014. PMID 23669268
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Ilyas S, Symons J, Bradley WP, Segal R, Taylor H, Lee K, Balkin M, Bain C, Ng I. A prospective randomised controlled trial comparing tracheal intubation plus manual in-line stabilisation of the cervical spine using the Macintosh laryngoscope vs the McGrath((R)) Series 5 videolaryngoscope. Anaesthesia. 2014 Dec;69(12):1345-50. doi: 10.1111/anae.12804. Epub 2014 Aug 2. PMID 25087907
- [Background] Hsu HT, Chou SH, Wu PJ, Tseng KY, Kuo YW, Chou CY, Cheng KI. Comparison of the GlideScope(R) videolaryngoscope and the Macintosh laryngoscope for double-lumen tube intubation. Anaesthesia. 2012 Apr;67(4):411-5. doi: 10.1111/j.1365-2044.2011.07049.x. Epub 2012 Feb 11. PMID 22324297
- [Background] Komatsu R, Kamata K, Sessler DI, Ozaki M. Airway scope and Macintosh laryngoscope for tracheal intubation in patients lying on the ground. Anesth Analg. 2010 Aug;111(2):427-31. doi: 10.1213/ANE.0b013e3181e3dfd2. Epub 2010 Jun 7. PMID 20529982
- [Background] Lin W, Li H, Liu W, Cao L, Tan H, Zhong Z. A randomised trial comparing the CEL-100 videolaryngoscope(TM) with the Macintosh laryngoscope blade for insertion of double-lumen tubes. Anaesthesia. 2012 Jul;67(7):771-6. doi: 10.1111/j.1365-2044.2012.07137.x. Epub 2012 Apr 30. PMID 22540996
- [Background] Mourao J, Moreira J, Barbosa J, Carvalho J, Tavares J. Soft tissue injuries after direct laryngoscopy. J Clin Anesth. 2015 Dec;27(8):668-71. doi: 10.1016/j.jclinane.2015.07.009. Epub 2015 Sep 26. PMID 26391674
- [Background] Lewis SR, Butler AR, Parker J, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011136. doi: 10.1002/14651858.CD011136.pub2. PMID 27844477
- [Background] Reynolds SF, Heffner J. Airway management of the critically ill patient: rapid-sequence intubation. Chest. 2005 Apr;127(4):1397-412. doi: 10.1378/chest.127.4.1397. PMID 15821222
- [Background] Di Marco P, Scattoni L, Spinoglio A, Luzi M, Canneti A, Pietropaoli P, Reale C. Learning curves of the Airtraq and the Macintosh laryngoscopes for tracheal intubation by novice laryngoscopists: a clinical study. Anesth Analg. 2011 Jan;112(1):122-5. doi: 10.1213/ANE.0b013e3182005ef0. Epub 2010 Nov 3. PMID 21048093
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Guimaraes-Pereira L, Costa M, Sousa G, Abelha F. Quality of recovery after anaesthesia measured with QoR-40: a prospective observational study. Braz J Anesthesiol. 2016 Jul-Aug;66(4):369-75. doi: 10.1016/j.bjane.2014.11.010. Epub 2015 Oct 20. PMID 27343786
- [Background] Sveinsdottir H, Borgthorsdottir T, Asgeirsdottir MT, Albertsdottir K, Asmundsdottir LB. Recovery After Same-Day Surgery in Patients Receiving General Anesthesia: A Cohort Study Using the Quality of Recovery-40 Questionnaire. J Perianesth Nurs. 2016 Dec;31(6):475-484. doi: 10.1016/j.jopan.2015.07.003. Epub 2016 May 5. PMID 27931699
- [Background] Invima - Instituto Nacional de Vigilancia de Medicamentos y Alimentos., Ministerio de Protección Social. Resolución No. 8430 del 4 de Octubre de 1993 - Por la cual se establecen las normas científicas, técnicas y administrativas para la investigación en salud. [Internet]. [cited 2017 Jan 20]. Available from: https://www.invima.gov.co/resoluciones-medicamentos/2977-resolucion-no-8430-del-4-de-octubre-de-1993.html
- [Background] La MDE, Social P. Ministerio De La Proteccion Social Resolucion número 2378 De 2008. 2008;2004(1271):1-10.
- [Background] Humanidades D De, Apartado B, España P. Universidad de Navarra Centro de Documentación de Bioética Declaración de Helsinki de la AMM - Principios éticos para las investigaciones médicas en seres humanos. 2013;1-8
- [Background] Favaloro A. Pautas éticas internacionales para la investigación biomédica en seres humanos [Internet]. Index Infectológico. 2008. 1-119 p. Available from: http://www.gramonbago.com.uy/imgnoticias/16791.pdf#page=11
- [Background] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955
- [Result] Richard M. Levitan M, Scott D. Cook-Sather M, E. Andrew Ochroch M. Demystifying Direct Laryngoscopy and Intubation. Hosp Physician [Internet]. 2000;1(59):47-56. Available from: http://w.hospitalphysician.com/pdf/hp_may00_intub.pdf